CLINICAL TRIAL: NCT02752139
Title: Cerebral Hemodynamics in Sleep Disorders
Status: Completed | Type: Observational
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: CHSD-01-R
Record Dates: First submitted 2016-03-07; First posted 2016-04-26 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Sleep Disorders, Intrinsic
Keywords: Sleep Disorders; Cerebral Hemodynamics; Dynamic Cerebral Auto-Regulation; Stroke
MeSH Terms: conditions — Sleep Disorders, Intrinsic; Sleep Wake Disorders; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients with sleep disorders
- normal individuals without sleep disorders

SUMMARY:
The purpose of this study is to determine the relationship between sleep disorders and cerebral hemodynamics.

DETAILED DESCRIPTION:
Sleep disorders continue to be the most unrecognized modifiable risk factor for stroke. The relationship between sleep disorders and vascular risk factors and stroke has been well-documented but not fully understood. The investigators hypothesize hemodynamics impairment to be its potential mechanism. It has been reported that sleep-related breathing disorder, a type of sleep disorders, contributed as a risk factor for stroke through hemodynamic and hematologic changes. The purpose of this study is to determine the relationship between different kind of sleep disorders and cerebral hemodynamics, including OSHAS, RLS, RBD, narcolepsy, etc. The dynamic cerebral auto-regulation (dCA) and Transcranial Doppler (TCD) will be used to evaluate cerebral hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* patients with sleep disorders
* meet the Diagnostic Criteria for Sleep Dyssomnias
* sufficient bilateral temporal bone windows for insonation of the MCA

Exclusion Criteria:

* middle cerebral artery (MCA) and/or other intracranial and/or extracranial major vascular 4 stenosis/occlusion, as diagnosed by a transcranial Doppler
* having a prior symptomatic cerebral vascular disease
* current arrhythmia, hyperthyroidism, anemia and unstable blood pressure, which may undermine hemodynamic stability
* inability to cooperate sufficiently to complete the dCA examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators conducted a prospective study of consecutive patients with sleep disorders treated at the Department of Neurology, First Hospital of Jilin University, China, from March 2016 to March 2017. Each patient was diagnosed with intrinsic sleep disorders by two neurologists according to the Diagnostic Criteria for Sleep Dyssomnias.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-05; Primary Completion 2018-08 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
phase difference(PD) in degree | 6 months
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.
the rate of recovery of cerebral blood flow velocity | 6 months
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.The details are same as outcome 1
gain in cm/s/mmHg | 6 months
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.The details are same as outcome 1

SECONDARY OUTCOMES:
mean MCA blood flow velocity (mCBFV) changes from supine to upright position | 6 months
pulsatility index (PI) changes from supine to upright position | 6 months
resistance index (RI) changes from supine to upright position | 6 months

OTHER OUTCOMES:
scores of Pittsburgh sleep quality index(PSQI) | 6 months
scores of Hamilton Anxiety Scale(HAMA) | 6 months
scores of Hamilton Depression Scale(HAMD) | 6 months
Polysomnography（PSG） | within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Deng F, Zhang Y, Zhang R, Tang Q, Guo Z, Lv Y, Wang Z, Yang Y. Compromised Dynamic Cerebral Autoregulation in Patients With Central Disorders of Hypersomnolence. Front Neurol. 2021 Mar 11;12:634660. doi: 10.3389/fneur.2021.634660. eCollection 2021. PMID 33776891